CLINICAL TRIAL: NCT01157156
Title: A Phase I, Multi-Center, Open Label, Safety and Tolerability Study of Single and Repeated Administrations of Escalating Dose(s) of NV1FGF Administered by Intra-Muscular Injection in Patients With Severe Peripheral Artery Occlusive Disease
Brief Title: Safety and Tolerability of NV1FGF in Patients With Severe Peripheral Artery Occlusive Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED10106; PM101 (Other: Gencell)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: XRP0038 (NV1FGF) — Pharmaceutical form:solution
  Route of administration: intramuscular

SUMMARY:
The primary objective is to evaluate safety and tolerability of single and repeated administrations of escalating doses of NV1FGF administered intramuscularly in patients with severe Peripheral Artery Occlusive Disease (PAOD), (Rutherford's Grade II, category 4 or Grade III, category 5 and 6).

Secondary objectives are:

* To determine the biological activity of NV1FGF on collateral artery development.
* To evaluate the activity of NV1FGF on hemodynamic and clinical parameters.

DETAILED DESCRIPTION:
Screening period of 30 days before dosing. Patients receive a single administration or repeated (2) administrations (with a 2-week interval) of NV1FGF. Patients are then followed for a period of 6 months

ELIGIBILITY:
Inclusion criteria:

* Severe PAOD defined as Rutherford's Grade II, category 4 or Grade III, category 5 and 6
* Pain at rest for at least 2 weeks duration and/or trophic lesions for at least the previous 14 days with no signs of healing (no reduction in ulcer size or depth)
* Objective evidence of peripheral vascular disease (resting Ankle Brachial Index < 0.4 and/or resting Toe Brachial Index < 0.3 and/or metatarsal Peripheral Vascular Resistance flat or barely pulsatile in the diseased limb on 2 consecutive examinations performed at least 2 weeks apart)
* Angiographic demonstration of total occlusion of the affected limb of one or more of the iliac, superficial femoral, popliteal and/or one or more infrapopliteal arteries
* Poor candidate for surgical intervention or revascularization procedures (no tibial artery incontinuity as defined from mid-leg distance from the foot and no autologous tissue available)

Exclusion criteria :

* Previous or current history of malignant disease. Patients who had successful tumor resection more than 10 years prior to inclusion into the study and had no recurrence and patients who had curatively resected basal/squamous cancer of the skin were allowed for inclusion
* Abnormal chest X-ray with suspected malignant tumor presence
* Positive stool hemoccult (expect if due to hemorrhoids)
* Positive Prostate Specific Antigen for men with suspected malignant tumor presence
* Abnormal mammography for women with suspected malignant tumor presence
* Papanicolaou smear (for women) of Class IV or Class V characterization
* Proliferative retinopathy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1999-06; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Safety assessment (adverse events, physical examination,vital signs,ECG, laboratory tests...) | 12 weeks

SECONDARY OUTCOMES:
hemodynamic parameters (TcPO2, Ankle Brachial Index, Toe Brachial Index, pulse volume recording) and angiography | 12 weeks
ulcers healing assessment (length, width, type, depth) | 12 weeks
pain assessment (self-administered visual analog scale) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development Study Director, Study Director — Sanofi
Locations (2):
- Minneapolis, Minnesota, United States
- Tempere, Finland

REFERENCES:
- [Derived] Niebuhr A, Henry T, Goldman J, Baumgartner I, van Belle E, Gerss J, Hirsch AT, Nikol S. Long-term safety of intramuscular gene transfer of non-viral FGF1 for peripheral artery disease. Gene Ther. 2012 Mar;19(3):264-70. doi: 10.1038/gt.2011.85. Epub 2011 Jun 30. PMID 21716303